CLINICAL TRIAL: NCT03258619
Title: Natriuresis as a Predictor of the Haemodynamic Response to Steroid Replacement Therapy in Patients in Septic Shock
Acronym: NARCOSE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Bouhemad-Nguyen 2016
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Aldosterone; Natriuresis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Aldosterone / renin dosage — Plasma levels of aldosterone and renin
Biological: Natriuresis — natriuresis levels

SUMMARY:
Septic shock is responsible in 20% of cases of acute adrenal insufficiency and in 50% of cases of chronic 'slow' adrenal insufficiency. Given the unpredictable nature of the response to the ACTH stimulation test, it is recommended to systematically start steroid replacement therapy with hydrocortisone hemisuccinate (HCHS) in patients in septic shock who do not respond to fluid resuscitation and who continue to suffer from haemodynamic instability despite increasing doses of noradrenaline.

The interest of this corticosteroid therapy lies in its ability to reduce the duration of treatment with catecholamines, though the results are conflicting with regard to an eventual benefit for mortality.

Steroid replacement therapy may be deleterious. It may increase the risk of sepsis and secondary septic shock. It is also implicated in critical-illness polyneuropathy and blood glucose dysregulation.

Today, there is no way to identify a population of patients who respond to corticosteroid therapy.

From a pathophysiological viewpoint, HCHS, as well as its glucocorticoid effects, may also exert mineralocorticoid effects able to compensate for the impaired renin angiotensin aldosterone system (RAAS), which is responsible for the refractory aspects of septic shock.

This hyperreninism-hypoaldosteronism is found with a prevalence of around 50% of cases and is defined by a plasma aldosterone/ plasma renin ratio < 2. It is associated with natriuresis >30 mmol/l.

We hypothesise that natriuresis > 30 mmol/l will make it possible to identify patients who respond to steroid replacement therapy in terms of catecholamine use.

ELIGIBILITY:
Inclusion Criteria:

* persons who have consented to take part
* Patients aged 18 to 85 years
* Admitted to an ICU for a first episode of septic shock
* With a dose of noradrenaline ≥ 0.25µg/kg/min
* Undergoing treatment with Hydrocortisone Hemisuccinate (HCHS)

Exclusion Criteria:

* Adult under guardianship
* Patients without national health insurance cover
* Pregnant or breast-feeding women
* Immunodepression (AIDS, corticosteroid treatment > 3 weeks, Organ graft, treatment with immunosuppressants)
* Recent intake of diuretics (< 6 h)
* Long-term ACE inhibitors or ARAII
* Chronic kidney failure (clearance < 60)
* Cirrhosis Child ≥ B
* Chronic heart failure (NYHA III and IV)
* Decision to limit or to stop treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalised for septic shock
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Variation in doses of noradrenaline | Day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France